CLINICAL TRIAL: NCT05964387
Title: Effect of Silver Diamine Fluoride on Local Anesthesia Efficacy in Molar Incisor Hypomineralization-affected Molars in Children: A Randomized Clinical Trial
Brief Title: Effect of Silver Diamine Fluoride on Local Anesthesia in Hypomineralized Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James R. Boynton, Clinical Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00228059
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Molar Incisor Hypomineralization; Anesthesia, Local
Keywords: Silver diamine fluoride
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: Subjects randomized for application of 38% silver diamine fluoride or placebo on hypomineralized permanent molar two weeks before operative dentistry.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject, care provider/outcomes assessor, and investigator will be blinded to which arm the tooth is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SDF (Experimental): 38% SDF applied to hypomineralized permanent molar two weeks prior to restorative care of the tooth.
  Interventions: Device: SDF
- Placebo (Placebo Comparator): Inert liquid (colored water) applied to hypomineralized permanent molar two weeks prior to restorative care of the tooth.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: SDF — 38% SDF will be applied to the hypoplastic area of the enrolled first permanent molar.
  Arms: SDF
Device: Placebo — An inert liquid will be applied to the hypoplastic area of the enrolled first permanent molar.
  Arms: Placebo

SUMMARY:
The purpose of this randomized, controlled clinical study is to evaluate if application of 38% SDF increases the efficacy of local anesthesia during operative dentistry on permanent molars affected by molar-incisor hypoplasia (MIH). The goal is to determine if pre-operative application of SDF results in improved local anesthesia and decrease in procedural pain in MIH affected teeth, thereby addressing an important challenge in routine clinical practice and contributing to the development of a treatment protocol for MIH affected molars.

DETAILED DESCRIPTION:
Molar incisor hypomineralization (MIH) is defined as a qualitative enamel defect of unknown etiology that affects one or more permanent molars and may also affect the permanent incisors. Clinically, the presentation of MIH depends on severity: lesions can range from mild, with white to yellow-brown discolored opacities, to severe, with extensive post-eruptive enamel breakdown and atypical caries. Hypomineralized enamel has increased porosity with reduced mineral content, which promotes bacteria penetration, resulting in development and rapid progression of dental caries and subclinical chronic pulp inflammation.

Treatment of teeth affected by MIH pose a clinical challenge due to several reasons. Post-eruptive breakdown of inadequately formed enamel exposes underlying dentin, resulting in hypersensitivity to hot and cold temperatures, air, and water. This increased tooth sensitivity leads to poor oral hygiene and subsequent plaque retention. Additionally, chronic subclinical inflammation of the pulp hypersensitizes the gamma-aminobutyric acid (GABA) receptors in the pulp nerve tissue and reduces the pain threshold in these teeth. This weakens the action of local anesthetics making it difficult to achieve adequate pain control during dental treatment.

Recently, 38% silver diamine fluoride (SDF), a solution of silver fluoride and ammonium ions, has been shown to be effective in tooth desensitization by blocking dentinal tubules and promoting remineralization of demineralized tooth structure. SDF can be useful in managing symptomatic MIH-affected teeth by stimulating the production of calcium fluoride and silver iodide, both of which are able to occlude dentinal tubules and reduce their patency.

The purpose of this randomized, controlled clinical study is to evaluate the efficacy of local anesthesia on MIH-affected molars treated with 38% SDF. The goal is to determine if pre-operative application of SDF results in improved local anesthesia and decrease in procedural pain in MIH affected teeth, thereby addressing an important challenge in routine clinical practice and contributing to the development of a treatment protocol for MIH affected molars.

ELIGIBILITY:
Inclusion Criteria:

* At least one hypomineralized first permanent molar with a primary cavitated caries lesion(s) or a cavitated tooth defect requiring restorative dental care with local anesthesia
* American Society of Anesthesiologists (ASA) Physical Status Classification I or II (healthy children or those with mild systemic disease)
* English speaking
* Subjects for which basic behavior guidance (non-pharmacological or nitrous oxide/oxygen) is indicated

Exclusion Criteria:

* Teeth with irreversible pulpitis and pulp necrosis
* Patients requiring advanced behavior management such as moderate sedation, general anesthesia, and/or active or passive restraint
* Inability of the child to cooperate due to special needs or other conditions
* Allergy to SDF, local anesthetic or other material component
* Subjects with ulcerative gingivitis or stomatitis
* Subjects with known sensitivity to silver or other heavy-metal ions
* Subjects showing abnormal skin sensitization in daily circumstances

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sixou and Barbosa-Rogier scale for local anesthesia efficacy | At least two weeks following application of SDF or placebo on the enrolled tooth
  Four point scale evaluating efficacy of local anesthesia

SECONDARY OUTCOMES:
Schiff Cold Air Sensitivity Scale | At least two weeks following application of SDF or placebo on the enrolled tooth
  Four point scale evaluating tooth sensitivity to cold

OTHER OUTCOMES:
Face, Legs, Activity, Cry, Consolability (FLACC) Scale | At least two weeks following application of SDF or placebo on the enrolled tooth
  Three point scale evaluating five components of behavior and expression of discomfort in children

CONTACTS AND LOCATIONS:
Overall Officials: James Boynton, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) is not planned to be shared.